CLINICAL TRIAL: NCT06835244
Title: Diagnostic Performance of PET/CT-PSMA in Patients With Non-prostatic PSMA-expressing Neoplasms: A Monocentric Observational Experience
Brief Title: Diagnostic Performance of PET/CT-PSMA in Patients With Non-prostatic PSMA-expressing Neoplasms
Acronym: MORE-PSMA
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MORE - PSMA
Record Dates: First submitted 2025-01-28; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: PSMA Positive Tumors or Tumor Tissues; Cancer
Keywords: PSMA PET/CT; PSMA expressing tumors
MeSH Terms: conditions — Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MORE PSMA POPULATION: Patients with tumors other than prostate cancer who may express PSMA
  Interventions: Other: 68Ga-PSMA-11

INTERVENTIONS:
Other: 68Ga-PSMA-11 — All patients with non prostatic neoplasm expressing PSMA undergo 68[Ga]Ga-PSMA-11-PET/CT
  Other Names: PSMA PET/CT

SUMMARY:
Study to collect data from PET/CT-PSMA performed in patients with neoplasms expressing PSMA, other than prostate cancer.

Objectives The primary objective is to evaluate the diagnostic performance of PET/CT-PSMA in the staging and management of patients with non-prostatic neoplasms expressing PSMA.

The secondary objective is to analyze the prognostic value of PET-PSMA in such neoplasms and the possible use in the selection of patients eligible for target therapies against neovascularization (i.e. monoclonal anti-VEGF antibodies) and radiopharmaceutical treatments (i.e. 177Lu-PSMA).

DETAILED DESCRIPTION:
Purpose of the register: This single-centre observational register is intended to collect data from PET/CT-PSMA performed in patients with neoplasms expressing PSMA, other than prostate cancer.

Design of the register: observational, pharmacological, non-profit, prospective, monocentric.

Duration of the record: The expected duration for the collection of PET/CT-PSMA examinations is 10 years.

Objectives The primary objective of the following registry is to evaluate the diagnostic performance of PET/CT-PSMA in the staging and management of patients with non-prostatic neoplasms expressing PSMA.

The secondary objective is to analyze the prognostic value of PET-PSMA in such neoplasms and the possible use in the selection of patients eligible for target therapies against neovascularization (i.e. monoclonal anti-VEGF antibodies) and radiopharmaceutical treatments (i.e. 177Lu-PSMA).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a neoplasm other than prostate carcinoma who are referred to our unit as part of the standard care pathway to undergo a PSMA PET/CT scan for staging, restaging, and pre- and post-treatment evaluation
* Signed informed consent for the collection and processing of data
* Minimum age 18 years old."

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with neoplasms other than prostate carcinoma, referred to the Nuclear Medicine Unit to undergo a PET/CT scan with PSMA.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
PSMA PET/CT performance | From the enrollment up to 10 years
  the evaluation of diagnostic performance of PSMA PET/CT and the positivity rate (%) globally and stratified by specific pathology in staging, re-staging and management of patients with non-prostatic neoplasms expressing PSMA.

SECONDARY OUTCOMES:
Prognostic and predictive value | From the enrollment up to 10 years
  Prognostic and predictive values (%) of PSMA PET/CT in such cancers and the possible use in the selection of patients eligible for target therapies against neovascularization and radioligand treatment according to specific score of PSMA expressing cells (%).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Farolfi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Nuclear Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided